CLINICAL TRIAL: NCT01241708
Title: Tandem Autologous Hematopoietic Stem Cell Transplant With Melphalan Followed by Melphalan and Bortezomib in Patients With Multiple Myeloma
Brief Title: Tandem Auto Stem Cell Transplant With Melphalan Followed by Melphalan and Bortezomib in Patients With Multiple Myeloma
Acronym: (Mel/MelVel)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001295; NCT01374958 (obsolete NCT alias)
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Auto Stem Cell Transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tandem Transplantation with Melphalan and Bortezomib (Experimental): Tandem autologous hematopoietic stem cell transplantation with melphalan followed by melphalan and bortezomib in patients with multiple myeloma
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.6mg/m2 on day -4 and day -1
  Other Names: Velcade

SUMMARY:
High dose chemotherapy with stem cell transplantation is commonplace in the treatment of multiple myeloma. This treatment uses a chemotherapy drug called Melphalan that has been used in several thousand bone marrow transplant recipients worldwide for the same or similar disorders.

DETAILED DESCRIPTION:
Many patients with multiple myeloma receive 2 stem cell transplantations within a few months of each other as part of their treatment. Usually the drug Melphalan is used for both transplants.

Bortezomib is a drug that is used for treating multiple myeloma and has been used in combination with melphalan for stem cell transplantation for patients with multiple myeloma.

The purpose of this trial is to study the effects of doing 2 transplants, first using melphalan and second using melphalan and bortezomib. The trial is aiming to find out if adding the Bortezomib to the second transplant will increase the chances of staying in remission longer.

ELIGIBILITY:
Changed from: Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma with either Durie-Salmon stage I, II, or III or ISS stage I, II or III, less than 12 months since initiation of systemic therapy
* ≥8x106 CD34+cells/kg available in cryopreservation in aliquots appropriate for tandem transplants
* Age: 18-75 years at time of transplantation
* KPS 70-100%
* Recovery from complications of prior therapies
* Gender: There is no gender restriction

Exclusion Criteria:

* Diagnosis other than multiple myeloma
* Chemotherapy or radiotherapy within 8 days of initiating treatment in this study
* Prior autologous or allogeneic transplantation (except as enrolled into this study)
* Uncontrolled bacterial, viral, fungal or parasitic infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2010-04-08 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Donato, MD, Principal Investigator — John Theurer Cancer Center at Hackensack University Medical Center
Locations (1):
- John Theurer Cancer Center @ Hackensack University Medical Center, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Adams J, Palombella VJ, Sausville EA, Johnson J, Destree A, Lazarus DD, Maas J, Pien CS, Prakash S, Elliott PJ. Proteasome inhibitors: a novel class of potent and effective antitumor agents. Cancer Res. 1999 Jun 1;59(11):2615-22. PMID 10363983
- [Background] Aghajanian C, Dizon DS, Sabbatini P, Raizer JJ, Dupont J, Spriggs DR. Phase I trial of bortezomib and carboplatin in recurrent ovarian or primary peritoneal cancer. J Clin Oncol. 2005 Sep 1;23(25):5943-9. doi: 10.1200/JCO.2005.16.006. PMID 16135465
- [Background] Alexanian R, Dimopoulos M. The treatment of multiple myeloma. N Engl J Med. 1994 Feb 17;330(7):484-9. doi: 10.1056/NEJM199402173300709. No abstract available. PMID 8289856
- [Background] Attal M, Huguet F, Schlaifer D, Payen C, Laroche M, Fournie B, Mazieres B, Pris J, Laurent G. Intensive combined therapy for previously untreated aggressive myeloma. Blood. 1992 Mar 1;79(5):1130-6. PMID 1536941
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495
- [Background] Attal M, Harousseau JL, Facon T, Guilhot F, Doyen C, Fuzibet JG, Monconduit M, Hulin C, Caillot D, Bouabdallah R, Voillat L, Sotto JJ, Grosbois B, Bataille R; InterGroupe Francophone du Myelome. Single versus double autologous stem-cell transplantation for multiple myeloma. N Engl J Med. 2003 Dec 25;349(26):2495-502. doi: 10.1056/NEJMoa032290. PMID 14695409
- [Background] Badros A, Barlogie B, Siegel E, Roberts J, Langmaid C, Zangari M, Desikan R, Shaver MJ, Fassas A, McConnell S, Muwalla F, Barri Y, Anaissie E, Munshi N, Tricot G. Results of autologous stem cell transplant in multiple myeloma patients with renal failure. Br J Haematol. 2001 Sep;114(4):822-9. doi: 10.1046/j.1365-2141.2001.03033.x. PMID 11564069
- [Background] Barlogie B, Jagannath S, Vesole DH, Naucke S, Cheson B, Mattox S, Bracy D, Salmon S, Jacobson J, Crowley J, Tricot G. Superiority of tandem autologous transplantation over standard therapy for previously untreated multiple myeloma. Blood. 1997 Feb 1;89(3):789-93. PMID 9028309
- [Background] Barlogie B, Kyle RA, Anderson KC, Greipp PR, Lazarus HM, Hurd DD, McCoy J, Moore DF Jr, Dakhil SR, Lanier KS, Chapman RA, Cromer JN, Salmon SE, Durie B, Crowley JC. Standard chemotherapy compared with high-dose chemoradiotherapy for multiple myeloma: final results of phase III US Intergroup Trial S9321. J Clin Oncol. 2006 Feb 20;24(6):929-36. doi: 10.1200/JCO.2005.04.5807. Epub 2006 Jan 23. PMID 16432076
- [Background] Berenson JR, Yang HH, Sadler K, Jarutirasarn SG, Vescio RA, Mapes R, Purner M, Lee SP, Wilson J, Morrison B, Adams J, Schenkein D, Swift R. Phase I/II trial assessing bortezomib and melphalan combination therapy for the treatment of patients with relapsed or refractory multiple myeloma. J Clin Oncol. 2006 Feb 20;24(6):937-44. doi: 10.1200/JCO.2005.03.2383. Epub 2006 Jan 17. PMID 16418495
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Blade J, Rosinol L, Sureda A, Ribera JM, Diaz-Mediavilla J, Garcia-Larana J, Mateos MV, Palomera L, Fernandez-Calvo J, Marti JM, Giraldo P, Carbonell F, Callis M, Trujillo J, Gardella S, Moro MJ, Barez A, Soler A, Font L, Fontanillas M, San Miguel J; Programa para el Estudio de la Terapeutica en Hemopatia Maligna (PETHEMA). High-dose therapy intensification compared with continued standard chemotherapy in multiple myeloma patients responding to the initial chemotherapy: long-term results from a prospective randomized trial from the Spanish cooperative group PETHEMA. Blood. 2005 Dec 1;106(12):3755-9. doi: 10.1182/blood-2005-03-1301. Epub 2005 Aug 16. PMID 16105975
- [Background] Child JA, Morgan GJ, Davies FE, Owen RG, Bell SE, Hawkins K, Brown J, Drayson MT, Selby PJ; Medical Research Council Adult Leukaemia Working Party. High-dose chemotherapy with hematopoietic stem-cell rescue for multiple myeloma. N Engl J Med. 2003 May 8;348(19):1875-83. doi: 10.1056/NEJMoa022340. PMID 12736280
- [Background] Cleveland, WS: Robust locally-weighted regression and smoothing scatterplots. J. Am Stat Assoc. 1979; 74: 829-836
- [Background] Cox, DR. Regression models and life tables (with discussion). J R Stat Soc B.1972; 34:187-220.
- [Background] Cusack JC Jr, Liu R, Houston M, Abendroth K, Elliott PJ, Adams J, Baldwin AS Jr. Enhanced chemosensitivity to CPT-11 with proteasome inhibitor PS-341: implications for systemic nuclear factor-kappaB inhibition. Cancer Res. 2001 May 1;61(9):3535-40. PMID 11325813
- [Background] Desikan R, Barlogie B, Sawyer J, Ayers D, Tricot G, Badros A, Zangari M, Munshi NC, Anaissie E, Spoon D, Siegel D, Jagannath S, Vesole D, Epstein J, Shaughnessy J, Fassas A, Lim S, Roberson P, Crowley J. Results of high-dose therapy for 1000 patients with multiple myeloma: durable complete remissions and superior survival in the absence of chromosome 13 abnormalities. Blood. 2000 Jun 15;95(12):4008-10. PMID 10845942
- [Background] Dixon DO, Simon R. Sample size considerations for studies comparing survival curves using historical controls. J Clin Epidemiol. 1988;41(12):1209-13. doi: 10.1016/0895-4356(88)90025-x. PMID 3062140
- [Background] Durie BG, Kyle RA, Belch A, Bensinger W, Blade J, Boccadoro M, Child JA, Comenzo R, Djulbegovic B, Fantl D, Gahrton G, Harousseau JL, Hungria V, Joshua D, Ludwig H, Mehta J, Morales AR, Morgan G, Nouel A, Oken M, Powles R, Roodman D, San Miguel J, Shimizu K, Singhal S, Sirohi B, Sonneveld P, Tricot G, Van Ness B; Scientific Advisors of the International Myeloma Foundation. Myeloma management guidelines: a consensus report from the Scientific Advisors of the International Myeloma Foundation. Hematol J. 2003;4(6):379-98. PMID 14671610
- [Background] Fassas AB, Barlogie B, Ward S, Jagannath S, Vesole D, Mattox S, Siegel D, Muwalla F, Zangari M, Anaissie E, Rhee FV, Thertulien R, Lee CK, Desikan R, Arzumanian V, McCoy J, Tricot G. Survival after relapse following tandem autotransplants in multiple myeloma patients: the University of Arkansas total therapy I experience. Br J Haematol. 2003 Nov;123(3):484-9. doi: 10.1046/j.1365-2141.2003.04646.x. PMID 14617011
- [Background] Fermand JP, Ravaud P, Chevret S, Divine M, Leblond V, Belanger C, Macro M, Pertuiset E, Dreyfus F, Mariette X, Boccacio C, Brouet JC. High-dose therapy and autologous peripheral blood stem cell transplantation in multiple myeloma: up-front or rescue treatment? Results of a multicenter sequential randomized clinical trial. Blood. 1998 Nov 1;92(9):3131-6. PMID 9787148
- [Background] Fermand JP, Katsahian S, Divine M, Leblond V, Dreyfus F, Macro M, Arnulf B, Royer B, Mariette X, Pertuiset E, Belanger C, Janvier M, Chevret S, Brouet JC, Ravaud P; Group Myelome-Autogreffe. High-dose therapy and autologous blood stem-cell transplantation compared with conventional treatment in myeloma patients aged 55 to 65 years: long-term results of a randomized control trial from the Group Myelome-Autogreffe. J Clin Oncol. 2005 Dec 20;23(36):9227-33. doi: 10.1200/JCO.2005.03.0551. Epub 2005 Nov 7. PMID 16275936
- [Background] Fonseca R, Barlogie B, Bataille R, Bastard C, Bergsagel PL, Chesi M, Davies FE, Drach J, Greipp PR, Kirsch IR, Kuehl WM, Hernandez JM, Minvielle S, Pilarski LM, Shaughnessy JD Jr, Stewart AK, Avet-Loiseau H. Genetics and cytogenetics of multiple myeloma: a workshop report. Cancer Res. 2004 Feb 15;64(4):1546-58. doi: 10.1158/0008-5472.can-03-2876. PMID 14989251
- [Background] Fossella FV, DeVore R, Kerr RN, Crawford J, Natale RR, Dunphy F, Kalman L, Miller V, Lee JS, Moore M, Gandara D, Karp D, Vokes E, Kris M, Kim Y, Gamza F, Hammershaimb L. Randomized phase III trial of docetaxel versus vinorelbine or ifosfamide in patients with advanced non-small-cell lung cancer previously treated with platinum-containing chemotherapy regimens. The TAX 320 Non-Small Cell Lung Cancer Study Group. J Clin Oncol. 2000 Jun;18(12):2354-62. doi: 10.1200/JCO.2000.18.12.2354. PMID 10856094
- [Background] Fossella F. Docetaxel + Cisplatin (DC) and Docetaxel + Carboplatin (DCb) vs Vinorelbine + Cisplatin (VC) in chemotherapy-naïve patients with advanced and metastatic non-small cell lung cancer (NSCLC): Results of a multicenter, randomized phase III study. European Journal of Cancer, European Cancer Conference, ECCO 11, 2001; Lisbon, Portugal. 37(suppl 6):S154. Abstract 562
- [Background] Gahrton G, Svensson H, Bjorkstrand B, Apperley J, Carlson K, Cavo M, Ferrant A, Fouillard L, Gratecos N, Gratwohl A, Guilhot F, Lambertenghi Deliliers G, Ljungman P, Masszi T, Milligan DW, Powles RL, Reiffers J, Samson JD, Stoppa AM, Vernant JP, Volin L, Wallvik J. Syngeneic transplantation in multiple myeloma - a case-matched comparison with autologous and allogeneic transplantation. European Group for Blood and Marrow Transplantation. Bone Marrow Transplant. 1999 Oct;24(7):741-5. doi: 10.1038/sj.bmt.1701975. PMID 10516677
- [Background] Goldberg SL, Klumpp TR, Magdalinski AJ, Mangan KF. Value of the pretransplant evaluation in predicting toxic day-100 mortality among blood stem-cell and bone marrow transplant recipients. J Clin Oncol. 1998 Dec;16(12):3796-802. doi: 10.1200/JCO.1998.16.12.3796. PMID 9850024
- [Background] Gouyette A, Hartmann O, Pico JL. Pharmacokinetics of high-dose melphalan in children and adults. Cancer Chemother Pharmacol. 1986;16(2):184-9. doi: 10.1007/BF00256174. PMID 3948304
- [Background] Hall AG, Tilby MJ. Mechanisms of action of, and modes of resistance to, alkylating agents used in the treatment of haematological malignancies. Blood Rev. 1992 Sep;6(3):163-73. doi: 10.1016/0268-960x(92)90028-o. PMID 1422285
- [Background] Harousseau JL, Attal M, Divine M, Marit G, Leblond V, Stoppa AM, Bourhis JH, Caillot D, Boasson M, Abgrall JF, et al. Autologous stem cell transplantation after first remission induction treatment in multiple myeloma: a report of the French Registry on autologous transplantation in multiple myeloma. Blood. 1995 Jun 1;85(11):3077-85. PMID 7756641
- [Background] Hideshima T, Richardson P, Chauhan D, Palombella VJ, Elliott PJ, Adams J, Anderson KC. The proteasome inhibitor PS-341 inhibits growth, induces apoptosis, and overcomes drug resistance in human multiple myeloma cells. Cancer Res. 2001 Apr 1;61(7):3071-6. PMID 11306489
- [Background] Hollmig K, Stover J, Talamo G, et al. Addition of bortezomib (Velcade™) to high dose melphalan (VelMel) as an effective conditioning regimen with autologous stem cell support in multiple myeloma (MM). Blood 2004;104:266a
- [Background] Jagannath S, Barlogie B, Berenson J, Siegel D, Irwin D, Richardson PG, Niesvizky R, Alexanian R, Limentani SA, Alsina M, Adams J, Kauffman M, Esseltine DL, Schenkein DP, Anderson KC. A phase 2 study of two doses of bortezomib in relapsed or refractory myeloma. Br J Haematol. 2004 Oct;127(2):165-72. doi: 10.1111/j.1365-2141.2004.05188.x. PMID 15461622
- [Background] Kergueris MF, Milpied N, Moreau P, Harousseau JL, Larousse C. Pharmacokinetics of high-dose melphalan in adults: influence of renal function. Anticancer Res. 1994 Nov-Dec;14(6A):2379-82. PMID 7825976
- [Background] LeBlanc R, Catley LP, Hideshima T, Lentzsch S, Mitsiades CS, Mitsiades N, Neuberg D, Goloubeva O, Pien CS, Adams J, Gupta D, Richardson PG, Munshi NC, Anderson KC. Proteasome inhibitor PS-341 inhibits human myeloma cell growth in vivo and prolongs survival in a murine model. Cancer Res. 2002 Sep 1;62(17):4996-5000. PMID 12208752
- [Background] Lee CK, Barlogie B, Zangari M, Fassas A, Anaissie E, Morris C, Van Rhee F, Cottler-Fox M, Thertulien R, Muwalla F, Mazher S, Badros A, Tricot G. Transplantation as salvage therapy for high-risk patients with myeloma in relapse. Bone Marrow Transplant. 2002 Dec;30(12):873-8. doi: 10.1038/sj.bmt.1703715. PMID 12476279
- [Background] Lightcap ES, McCormack TA, Pien CS, Chau V, Adams J, Elliott PJ. Proteasome inhibition measurements: clinical application. Clin Chem. 2000 May;46(5):673-83. PMID 10794750
- [Background] McElwain TJ, Powles RL. High-dose intravenous melphalan for plasma-cell leukaemia and myeloma. Lancet. 1983 Oct 8;2(8354):822-4. doi: 10.1016/s0140-6736(83)90739-0. PMID 6137651
- [Background] Mehta J, Tricot G, Jagannath S, Ayers D, Singhal S, Siegel D, Desikan K, Munshi N, Fassas A, Mattox S, Vesole D, Crowley J, Barlogie B. Salvage autologous or allogeneic transplantation for multiple myeloma refractory to or relapsing after a first-line autograft? Bone Marrow Transplant. 1998 May;21(9):887-92. doi: 10.1038/sj.bmt.1701208. PMID 9613780
- [Background] Mitsiades N, Mitsiades CS, Richardson PG, Poulaki V, Tai YT, Chauhan D, Fanourakis G, Gu X, Bailey C, Joseph M, Libermann TA, Schlossman R, Munshi NC, Hideshima T, Anderson KC. The proteasome inhibitor PS-341 potentiates sensitivity of multiple myeloma cells to conventional chemotherapeutic agents: therapeutic applications. Blood. 2003 Mar 15;101(6):2377-80. doi: 10.1182/blood-2002-06-1768. Epub 2002 Nov 7. PMID 12424198
- [Background] NATHANS D, FAHEY JL, POTTER M. The formation of myeloma protein by a mouse plasma cell tumor. J Exp Med. 1958 Jul 1;108(1):121-30. doi: 10.1084/jem.108.1.121. PMID 13549645
- [Background] Orlowski RZ, Stinchcombe TE, Mitchell BS, Shea TC, Baldwin AS, Stahl S, Adams J, Esseltine DL, Elliott PJ, Pien CS, Guerciolini R, Anderson JK, Depcik-Smith ND, Bhagat R, Lehman MJ, Novick SC, O'Connor OA, Soignet SL. Phase I trial of the proteasome inhibitor PS-341 in patients with refractory hematologic malignancies. J Clin Oncol. 2002 Nov 15;20(22):4420-7. doi: 10.1200/JCO.2002.01.133. PMID 12431963
- [Background] Orlowski RZ, Voorhees PM, Garcia RA, Hall MD, Kudrik FJ, Allred T, Johri AR, Jones PE, Ivanova A, Van Deventer HW, Gabriel DA, Shea TC, Mitchell BS, Adams J, Esseltine DL, Trehu EG, Green M, Lehman MJ, Natoli S, Collins JM, Lindley CM, Dees EC. Phase 1 trial of the proteasome inhibitor bortezomib and pegylated liposomal doxorubicin in patients with advanced hematologic malignancies. Blood. 2005 Apr 15;105(8):3058-65. doi: 10.1182/blood-2004-07-2911. Epub 2004 Dec 30. PMID 15626743
- [Background] Paccagnella A, Chiarion-Sileni V, Soesan M, Baggio G, Bolzonella S, De Besi P, Casara D, Frizzarin M, Salvagno L, Favaretto A, et al. Second and third responses to the same induction regimen in relapsing patients with multiple myeloma. Cancer. 1991 Sep 1;68(5):975-80. doi: 10.1002/1097-0142(19910901)68:53.0.co;2-o. PMID 1913491
- [Background] Palumbo A, Bringhen S, Petrucci MT, Musto P, Rossini F, Nunzi M, Lauta VM, Bergonzi C, Barbui A, Caravita T, Capaldi A, Pregno P, Guglielmelli T, Grasso M, Callea V, Bertola A, Cavallo F, Falco P, Rus C, Massaia M, Mandelli F, Carella AM, Pogliani E, Liberati AM, Dammacco F, Ciccone G, Boccadoro M. Intermediate-dose melphalan improves survival of myeloma patients aged 50 to 70: results of a randomized controlled trial. Blood. 2004 Nov 15;104(10):3052-7. doi: 10.1182/blood-2004-02-0408. Epub 2004 Jul 20. PMID 15265788
- [Background] Pandit S, Vesole DH. Relapsed multiple myeloma. Curr Treat Options Oncol. 2001 Jun;2(3):261-9. doi: 10.1007/s11864-001-0040-6. PMID 12057126
- [Background] Papandreou C, Daliani D, Millikan RE, Tu S, Pagliaro L, Adam J. Phase I Study of Intravenous (I.V.) Proteasome Inhibitor PS-341 in Patients (Pts) with Advanced Malignancies. Proc Am Soc Clin Oncol, 2001. Abstract 340
- [Background] Pineda-Roman M, Fox MH, Hollmig KA, et al. Retrospective analysis of fractionated high-dose melphalan (F-Mel) and bortezomib-thalidomide-dexamethasone (VTD) with autotransplant (AT) support for advanced and refractory multiple myeloma (AR-MM). Blood 2006;108:884a
- [Background] Pinguet F, Martel P, Fabbro M, Petit I, Canal P, Culine S, Astre C, Bressolle F. Pharmacokinetics of high-dose intravenous melphalan in patients undergoing peripheral blood hematopoietic progenitor-cell transplantation. Anticancer Res. 1997 Jan-Feb;17(1B):605-11. PMID 9066587
- [Background] Reece PA, Hill HS, Green RM, Morris RG, Dale BM, Kotasek D, Sage RE. Renal clearance and protein binding of melphalan in patients with cancer. Cancer Chemother Pharmacol. 1988;22(4):348-52. doi: 10.1007/BF00254244. PMID 3168148
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Richardson PG, Sonneveld P, Schuster MW, Irwin D, Stadtmauer EA, Facon T, Harousseau JL, Ben-Yehuda D, Lonial S, Goldschmidt H, Reece D, San-Miguel JF, Blade J, Boccadoro M, Cavenagh J, Dalton WS, Boral AL, Esseltine DL, Porter JB, Schenkein D, Anderson KC; Assessment of Proteasome Inhibition for Extending Remissions (APEX) Investigators. Bortezomib or high-dose dexamethasone for relapsed multiple myeloma. N Engl J Med. 2005 Jun 16;352(24):2487-98. doi: 10.1056/NEJMoa043445. PMID 15958804
- [Background] Richardson PG, Weller E, Jagannath S, Avigan DE, Alsina M, Schlossman RL, Mazumder A, Munshi NC, Ghobrial IM, Doss D, Warren DL, Lunde LE, McKenney M, Delaney C, Mitsiades CS, Hideshima T, Dalton W, Knight R, Esseltine DL, Anderson KC. Multicenter, phase I, dose-escalation trial of lenalidomide plus bortezomib for relapsed and relapsed/refractory multiple myeloma. J Clin Oncol. 2009 Dec 1;27(34):5713-9. doi: 10.1200/JCO.2009.22.2679. Epub 2009 Sep 28. PMID 19786667
- [Background] Rowley SD, Siegel, D, Donato ML,et al. Combination melphalan and bortezomib conditioning with autologous hematopoeitic stem cell support in patients with advanced multiple myeloma. A phase I/II study. Blood 2009;114:499
- [Background] Samuels BL, Bitran JD. High-dose intravenous melphalan: a review. J Clin Oncol. 1995 Jul;13(7):1786-99. doi: 10.1200/JCO.1995.13.7.1786. PMID 7602368
- [Background] Siegel DS, Desikan KR, Mehta J, Singhal S, Fassas A, Munshi N, Anaissie E, Naucke S, Ayers D, Spoon D, Vesole D, Tricot G, Barlogie B. Age is not a prognostic variable with autotransplants for multiple myeloma. Blood. 1999 Jan 1;93(1):51-4. PMID 9864145
- [Background] Spanswick VJ, Craddock C, Sekhar M, Mahendra P, Shankaranarayana P, Hughes RG, Hochhauser D, Hartley JA. Repair of DNA interstrand crosslinks as a mechanism of clinical resistance to melphalan in multiple myeloma. Blood. 2002 Jul 1;100(1):224-9. doi: 10.1182/blood.v100.1.224. PMID 12070031
- [Background] Teicher BA, Ara G, Herbst R, Palombella VJ, Adams J. The proteasome inhibitor PS-341 in cancer therapy. Clin Cancer Res. 1999 Sep;5(9):2638-45. PMID 10499643
- [Background] Tricot G, Jagannath S, Vesole DH, Crowley J, Barlogie B. Relapse of multiple myeloma after autologous transplantation: survival after salvage therapy. Bone Marrow Transplant. 1995 Jul;16(1):7-11. PMID 7581132
- [Background] Tricot G, Alberts DS, Johnson C, Roe DJ, Dorr RT, Bracy D, Vesole DH, Jagannath S, Meyers R, Barlogie B. Safety of autotransplants with high-dose melphalan in renal failure: a pharmacokinetic and toxicity study. Clin Cancer Res. 1996 Jun;2(6):947-52. PMID 9816255
- [Background] Tricot G, Spencer T, Sawyer J, Spoon D, Desikan R, Fassas A, Badros A, Zangari M, Munshi N, Anaissie E, Toor A, Barlogie B. Predicting long-term (> or = 5 years) event-free survival in multiple myeloma patients following planned tandem autotransplants. Br J Haematol. 2002 Jan;116(1):211-7. doi: 10.1046/j.1365-2141.2002.03231.x. PMID 11841419
- [Background] Vesole DH, Barlogie B, Jagannath S, Cheson B, Tricot G, Alexanian R, Crowley J. High-dose therapy for refractory multiple myeloma: improved prognosis with better supportive care and double transplants. Blood. 1994 Aug 1;84(3):950-6. PMID 7913845

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tandem Transplantation With Melphalan and Bortezomib
Started | 148
Completed | 92
Not Completed | 56
Not completed — Withdrawal by Subject | 6
Not completed — Screen Failure | 6
Not completed — Did not move forward with 2nd Transplant | 39
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Tandem Transplantation With Melphalan and Bortezomib
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 126
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years] | 56.4 [32.4 to 72.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 123
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 13
  White | 108
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Progression-free Survival of Patients With Multiple Myeloma Treated With Tandem Cycles of High-dose Melphalan Followed by High-dose Melphalan in Combination With Bortezomib With Autologous HSC Transplantation.
Description: Progression-free survival of participants that received tandem transplants on study
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Tandem Transplantation With Melphalan and Bortezomib
Number analyzed (Participants) | 94
Percent | 73.8 [64.3 to 82.2]

2. Secondary Outcome: To Determine the Response Rate of Patients With Multiple Myeloma Treated With High-dose Melphalan or High-dose Melphalan in Combination With Bortezomib Given in Tandem Transplants.
Description: Overall response rate of participants after completing tandem transplant. Overall Response rate defined as the composite endpoint of response to treatment which includes Complete Response (CR), Partial Response (PR), stable disease (SD) as defined in International Response Criteria.
Time Frame: 3 years
Population: 94 participant response assessed after completion of tandem transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Transplantation With Melphalan and Bortezomib
Number analyzed (Participants) | 94
Participants | 86

3. Secondary Outcome: To Determine the Overall Survival of Patients With Multiple Myeloma Treated With High-dose Melphalan or High-dose Melphalan in Combination With Bortezomib Given in Tandem Transplants.
Description: Survival rate of participants after completion of tandem transplant
Time Frame: 3 years
Population: 94 participant survival assessed after completion of tandem transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Tandem Transplantation With Melphalan and Bortezomib
Number analyzed (Participants) | 94
Participants | 76

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed for up to 3 years. Serious Adverse Events were assessed up to 100 days after bone marrow transplant
Description: SAEs are reported through 100 days after bone marrow transplant. Other (Not Including Serious) Adverse Events were not analyzed
Arm/Group | Tandem Transplantation With Melphalan and Bortezomib
All-Cause Mortality (participants affected / at risk) | 46/142
Serious Adverse Events (participants affected / at risk) | 67/142
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tandem Transplantation With Melphalan and Bortezomib (N=142)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Infection (Infections and infestations) | 15
Disease Progression (Investigations) | 26
Fever (Investigations) | 3
Engraftment Syndrome (Immune system disorders) | 4
Failure to Thrive (Investigations) | 2
RSV (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Perrirectal Abcess (Infections and infestations) | 1
Subdermal Hematoma (Vascular disorders) | 1
Acute Renal Insufficiency (Renal and urinary disorders) | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 1
CMV Viremia (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT01241708/Prot_SAP_000.pdf